CLINICAL TRIAL: NCT05247333
Title: Implementation, Integration and Sustainability of a Minor Ailment Service in Usual Practice of Community Pharmacy
Brief Title: Implementation of a Minor Ailment Service in Community Pharmacy Practice
Acronym: INDICA+PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Spanish Society of Community Pharmacy (Unknown); Pharmaceutical Association, Valencia (MICOF) (Unknown); Pharmaceutical Association, Madrid (Colegio Oficial de Farmacéuticos de Madrid) (Unknown); Pharmaceutical Association, Gipuzkoa (Colegio Oficial de Farmacéuticos de Gipuzkoa) (Unknown); Pharmaceutical Association, Málaga (Colegio Oficial de Farmacéuticos de Málaga) (Unknown); Pharmaceutical Association, Castellón (Colegio Oficial de Farmacéuticos de Castellón) (Unknown); Pharmaceutical Association of Valladolid (Colegio Oficial de Farmacéuticos de Valladolid) (Unknown)
Responsible Party: Principal Investigator, Noelia Amador Fernández, Project coordinator, Universidad de Granada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IndicaPROImp-2019-v2
Record Dates: First submitted 2021-12-01; First posted 2022-02-18 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Acne; Bites; Burns; Cold; Cold Sore Mouth; Constipation; Cough; Dental Trauma; Dermatitis; Diarrhea; Dry Eye; Dysmenorrhea; Flatulence; Foot Fungal Infection; Hemorrhoids; Headache; Heartburn; Hyperhidrosis; Mouth Ulcer; Musculoskeletal Pain; Nasal Congestion; Rash; Red Eye; Sleep Disorder; Soft Tissue Injuries; Sore Throat; Stress Disorder, Acute; Temperature Regulation Disorder; Vaginal Candidiasis; Varicose Veins; Vomiting
Keywords: Minor ailments
MeSH Terms: conditions — Acne Vulgaris; Bites and Stings; Burns; Common Cold; Constipation; Cough; Dermatitis; Diarrhea; Dry Eye Syndromes; Dysmenorrhea; Flatulence; Hemorrhoids; Headache; Heartburn; Hyperhidrosis; Oral Ulcer; Musculoskeletal Pain; Nasal Obstruction; Exanthema; Sleep Wake Disorders; Soft Tissue Injuries; Pharyngitis; Stress Disorders, Traumatic, Acute; Candidiasis, Vulvovaginal; Varicose Veins; Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients presenting with minor ailments or requesting a non-prescription product. (Experimental): Community pharmacists working with agreed protocols with primary care physicians respond to all type of patients presenting with minor ailments or requesting a non-prescription product.
  Following this consultation, patients are followed up after ten days.
  Interventions: Other: Minor ailment service

INTERVENTIONS:
Other: Minor ailment service — The service had several components: agreed standard operational procedures between community pharmacists and primary care physicians for 31 minor ailments, IT based consultation protocol and training before and during the study for the pharmacists. Practice change facilitators were used to confirm the fidelity of the intervention.

SUMMARY:
Self-care and self-medication are commonly the treatments of choice for the management of minor ailments. Minor ailments can be treated through community pharmacy using a Minor Ailment Service (MAS). The INDICA+PRO Impact Study, evaluated the clinical, economic and humanistic impact of a MAS, concluding that community pharmacies could greatly benefit the health system. Thus, the following objectives were defined for the INDICA+PRO implementation study.

The primary objective is to implement a standardised MAS in usual practice in community pharmacy in Spain. The secondary objectives include an evaluation of the clinical and economic outcomes and the role and impact of two different models of change agents. A pragmatic study with an effectiveness-implementation hybrid design type 3 will be undertaken using the Framework for the Implementation of Services in Pharmacy (FISpH). The study will be carried between October 2020 and December 2022. Two type of practice change facilitators FaFa and SEFaFa. Their main function, using the Observe-Plan-Do-Study-Act process, will be to facilitate the implementation through individualised continuous support to providers of the MAS. The depth and breadth of support to pharmacist providers by each type of change agents will vary.

Pharmaceutical Associations (PA) and/or Spanish Society of Community Pharmacy (SEFAC) will invite community pharmacies/pharmacists. Participating pharmacists will need to sign a commitment form. The second study population will consist of patients presenting with minor ailments or requesting a non-prescription medication. Recruitment of patients will be carried out by the pharmacist providers. The inclusion criteria will be: patients or caregivers (aged ≥18 years, or younger if they are accompanied by an adult) presenting with 31 minor ailments, grouped into five categories (respiratory, moderate pain, digestive, dermatological and other) with pre-agreed referral protocols. Other symptoms may be included at the discretion of the pharmacists. The exclusion criteria will be patients who do not provide informed consent.

The patient/pharmacist intervention will consist of a MAS protocol adapted for each symptom. The consultation will be record in an electronic data capture system (SEFAC eXPERT®-) that provides a step-by-step approach with protocols and clinical information embedded.

The FISpH model will be used to guide the implementation of MAS. Two types of change agents, FaFas and SeFaFas, previously trained for 18 hours, will be used to facilitate the implementation. During each of the stages (exploration, preparation, testing and operation, and initial sustainability), strategies will be used by FaFas and SeFaFas to moderate implementation factors. The impact of strategies will be evaluated. Data on pharmacy/pharmacist's provider performance and patient outcomes will be provided to pharmacist, change agents and PA and SEFAC. FaFas and SeFaFas will have a classification system for barriers and facilitators derived from the constructs in the Consolidated Framework for Implementation Research (CFIR). The classification system for implementation strategies consists of an adaptation of the facilitation activities listed by Dogherty et al. These will be documented in an electronic data capture system.

FaFas will train their pharmacists (max. of 25 pharmacies) for 6 hours and subsequently provide at least monthly follow-up.

The research team will provide ongoing feedback and support to the FaFas and SeFaFas through periodically, hold group meetings by video conference between the research group and all the FaFas and SeFaFas. The research group will provide formal reports on the implementation process and patient outcomes. Other forms of communication such as emails, telephone calls or WhatsApp messaging will also be available.

Implementation and patient consultation process and outcome variables will be measured such as reach, fidelity and integration. Outcome service indicators will be clinical, economic and humanistic. A patient follow up will occur at a maximum of 10 days. Continuous variables will be reported using mean and standard deviation, or median and percentiles. Categorical variables will be reported using percentages. T Student's test or the ANOVA test or Kruskal-Wallis. χ2 test, Fisher's exact test or Yate's chi-squared will also be used. To determine the relationship between the dependent and the independent variables, logistic regression models will be performed including the variables with statistical significance in the bivariate model. The level of significance will be set at p <0.05. Machine learning and big data techniques are being considered for predictive modelling.

The research team will only have access to de-identified data of pharmacists and patients. This study protocol has been approved by the Granada Research Ethics Committee on the 5th February 2020.

DETAILED DESCRIPTION:
INDICA+PRO Implementation Programme for the Implementation, Integration and Sustainability of a Standardised Minor Ailment Service in Usual Practice in Community Pharmacy

Background The World Health Organization (WHO) stated in 2009 that self-care is one of the essential components for achieving health objectives, as it directs and improves access to the appropriate level of healthcare system and reduces costs. Self-care and self-medication are commonly the treatments of choice for the management of minor ailments. Encouraging self-care promotes the improvement of the public's knowledge and skills to optimise decision-making related to health. Access to quality information at appropriate levels of health literacy is an essential element in the self-care process; and thus, health professionals, particularly community pharmacists, play a fundamental role.

Minor ailments are defined by Faus-Dáder et al. as "a health problem that is non-serious in nature, self-limited and of short duration, which has no relationship with the clinical manifestations of any other health problems suffered by the patient, or with the effects (desired or not) of any medication taken by the individual. Minor ailments do not require a medical diagnosis and respond to or are alleviated by symptomatic treatments".

Minor ailments can be treated through community pharmacy using a Minor Ailment Service (MAS). In Spain MAS was defined in 2019 by the "Pharmaceutical Care in Community Pharmacy Forum" (PC-CPF) as "the professional pharmaceutical service provided when a patient or caregiver visits a community pharmacy consulting a specific health problem and requesting the most appropriate remedy". PC-CPF includes a patient request for a non-prescription drug as part of a MAS. Responding to symptoms presented by patients and dealing with requests for non-prescription medication account for between 9% and 16% of the activity of community pharmacies. However, these activities are not legally classified as MAS.

A previous phase of the INDICA+PRO program, the INDICA+PRO Impact Study, evaluated for the first time in Spain the clinical, economic and humanistic impact of a MAS, concluding that community pharmacies could greatly benefit the health system through a more efficient treatment of minor ailments. In turn, increasing the accessibility of patients to the healthcare system as well as ensuring its future sustainability. Thus, the following objectives were defined for an implementation study.

Objectives Primary Objective To develop, implement and integrate a standardised MAS in usual practice in community pharmacy in Spain.

Secondary Objectives

* To evaluate the clinical outcomes of the standardised MAS in community pharmacy and compare these to the results obtained during the INDICA+PRO Impact Study Impact phase.
* To evaluate the role and impact of two different models of Change Agents: Pharmaceutical Facilitators (FaFas) and Pharmaceutical Facilitators of SEFAC (SeFaFas).

Method Research Design A pragmatic study with an effectiveness-implementation hybrid design type 3 using the Framework for the Implementation of Services in Pharmacy (FISpH).

Scope of study The study will be carried out in Spanish community pharmacies. The study will take place between October 2020 and December 2022.

Facilitation process of the MAS Traditional formal training is not an effective way to promote changes in behaviour or professional practice. Therefore, for this study, the ongoing support of Change Agents will be explored. These Change Agents will continuously monitor and assist in resolving barriers that appear during the implementation process and reinforce facilitators. Consequently, this study will evaluate the roles of the different models of Change Agents (FaFas and SeFaFas). FaFas are specifically trained pharmacists that promote change in professional practice and their main function is to intervene and facilitate this change through individualised continuous support and assistance to the pharmacist providers of the MAS. The FaFa is responsible for conducting on-site training and providing feedback and advice to the pharmacists, as well as being available by email, telephone, WhatsApp or video conference. FaFas will be employed by their participating Pharmaceutical Association. A SeFaFa is a "Spanish Society of Community Pharmacy" (SEFAC) member who volunteers to train and monitor participating pharmacies as well as participant in the study. The level of support provided is lower than that of the FaFas. Pharmacist providers can resolve queries with the SEFaFa via email, telephone, WhatsApp or video conference, however SeFaFas will not offer periodic follow-ups nor monthly on-site visits.

Throughout the cyclical, continuous and individualised facilitation process, the Change Agents will interact with their pharmacists and pharmacies to:

1. Identify implementation factors and prioritize them for action
2. Analyse the causes
3. Design individualised action (implementation strategies)
4. Study the impact of the strategy (s)
5. Redefine strategies based on feedback from the pharmacists and outcomes The process of facilitation is based on the PDSA cycle (Observe-Plan-Do-Study-Act), a method of continuous quality improvement designed to achieve sustainable change in practice through interventions and continuous evaluation.

Pharmaceutical Association (PA) and/or SEFAC will invite, through a number of channels, community pharmacies/pharmacists in selected study provinces to take part voluntarily. In the provinces where a PA is part of the study, the FaFa will be employed. All pharmacies will be invited by the PA by email. In provinces without a participating PA, a SEFaFa will be selected, and the invitation to participate will be made by SEFAC, also through an emailed invitation.

Pharmacies will have two weeks to decide whether to participate in the study. In provinces with participating PAs that have more than 25 pharmacies accepting the invitation, a random distribution into two groups will occur. The first group will consist of a maximum of 25 pharmacies and will be assigned to a FaFa. The second group will be assigned to a SEFaFa. In provinces with no participating PA, all pharmacies will be assigned to a SEFaFa. A maximum target of 1000 pharmacists have been set due to resource limitations. Only an intervention group will exist Participating pharmacist will need to sign a commitment form to be eligible to participate in the study.

Description of the pharmacist-patient intervention in the Standardised MAS

The patient /pharmacist intervention is described below. The generic MAS protocol was taken from the "Practical Guide for Pharmaceutical Care Services in the Community Pharmacy":

1. Patient Interview: the pharmacist will identify the patient and the reason for the consultation and whether any previous actions were carried out in an attempt to solve the symptoms, whether the patient is prescribed or is using any other medications and whether they have any allergies, intolerances or other concomitant diseases. If relevant, establish whether the patient is pregnant or breast feeding. The duration of the symptom will be determined.
2. Evaluation of the Information: identification of any existing referral criteria, drug-related problems (DRP) and/or negative outcomes associated with medication (NOM).
3. Action: the pharmacist provider can offer a non-prescription medication with the relevant information or a non-pharmacological treatment, which can be health education, hygienic-dietary measures or advice on healthy lifestyle habits. The pharmacist can also refer the patient to their primary care physician, to any other healthcare professional or for another pharmaceutical service.
4. Record in the Consultation in an Electronic Data Capture system - SEFAC eXPERT® IT system: the sex and age of the patient, the reason for the consultation, any previous actions that were carried out in an attempt to solve the symptoms, the proposed intervention and/or action (including any treatment offered, if applicable) and the outcome of the MAS.

Community pharmacists will carry out the intervention using symptom specific protocols that were previously agreed with primary care physicians. These protocols will include information on the minor ailment, referral criteria, prevention measures and possible treatments (both pharmacological and non-pharmacological). These symptom specific protocols are included in the SEFAC eXPERT® IT system.

Implementation Model of the Service To guide the implementation of MAS, the FISpH model will be used. This model proposes five different stages.

Implementation Stages

• Exploration: preparation of the pharmacy system and environment for the implementation of the MAS.

This exploration will include: system exploration with possible participants community pharmacist owners and providers who have been invited to participate, training of change agents and discussions with senior management at each of the PAs and SEFAC.

* Preparation: education and training of the owners of community pharmacies and their pharmacists. The training will include the fundamentals of implementation science and clinical protocols.
* Testing and operation: facilitation of the implementation of the MAS and promotion of its integration in the pharmacy using Change Agents. Feedback on testing process by change agents to providers. Data on pharmacy/pharmacist's provider performance and patient outcomes will be provided to pharmacist, change agents and PA and SEFAC.
* Initial sustainability: integration of the MAS into the pharmacy's daily practice and maintaining the continuity in its provision.

During each of the stages (exploration, preparation, testing and operation, and initial sustainability), implementation strategies will be used by FaFas and SeFaFas to assist moderate implementation factors (overcome barriers, promote facilitators and increase the use of the implementation process). Implementation factors (barriers and facilitators) will be grouped into five domains. The impact of any used strategies (grouped into four stages of facilitation) on the implementation factors will be evaluated.

Implementation Indicators

Evaluation throughout the different stages of the FISpH model will be carried out according to the following criteria:

* Exploration (considered as the number of pharmacists that wish to enrol in the study) and the percentage of pharmacies that accept the invitation to participate in the study.
* Preparation (considered as the number of pharmacies that complete the training to provide the Service and record between 1 - 4 consultations per month per pharmacist). The percentage of pharmacies that accept the invitation to participate and complete the initial implementation training will be calculated in relation to those that expressed their willingness to participate in the study.
* Testing: the percentage of pharmacies that complete the initial training implementation module for providers and undertake MAS with half of the target consultations (record 5 to 10 consultations per month per pharmacist).
* Implementation (considered as the number of pharmacies that perform the MAS on the full number of target patients): the percentage of pharmacies that perform the MAS on the full number of target patients will be calculated (11 or more consultations per month per pharmacist).
* Initial sustainability (considered as the number of pharmacies that recruit and complete the MAS for the full number of target consultations, 11 or more consultations per month for a further 6 months): the percentage of pharmacies that progress from the implementation stage to the initial sustainability stage will be calculated.

This data will be obtained directly from the SEFAC eXPERT® IT system. Training session for the Change Agents (FaFa and SEFaFa) There will be an 18-hour prior training for FaFas and a 12-hour session for SeFaFas, covering general concepts of the MAS, good practices of the MAS in Community Pharmacy, patient and interprofessional communication, data from the INDICA+PRO Impact study, protocols and primary physician referral criteria, SEFAC eXPERT® registration, case studies and the Implementation study protocol. FaFas and SeFaFas will receive ongoing training, at least one per month, on the characteristics and tasks of change facilitators, such as recognising barriers and facilitators, as well as designing the relevant implementation strategies.

Identification of Implementation Factors (barriers and facilitators) FaFas and SeFaFas will be provided with a classification system for barriers and facilitators that they will use as a tool to assist analyses when interacting with their pharmacies/pharmacists. These interactions/process will be documented in an Electronic Data Capture (EDC). The classification system consists of an adaptation of the constructs listed in the Consolidated Framework for Implementation Research (CFIR).

Design of implementation strategies FaFas and SeFaFas will be provided with a classification system for implementation strategies which they will use to design strategies and to document in the Electronic Data Capture (EDC). This classification system consists of an adaptation of the facilitation activities listed by Dogherty et al.

Training session for pharmacists in participating pharmacies

There will be two options for the pharmacist provider training:

1. FaFas will train their pharmacists (o a maximum of 25 pharmacies) and subsequently provide at least monthly follow-up.
2. SeFaFas will train their pharmacists without PA support. The participating pharmacists will be trained for an approximate period of 6 hours before the start of the study. The objective of these sessions will be to equip pharmacists with the necessary clinical knowledge and skills to carry out the MAS.

Competencies to be covered include the ability to:

* Implement MAS in accordance with the Good Practices in Community Pharmacy in Spain.
* Undertake minor ailment assessment and treatment, including the dispensing of appropriate non-prescription medications.
* Have communication techniques and skills for use with patients, physicians and other health care providers.
* Advice and provide information for patients on the use of non-prescription drugs.
* To have the knowledge to appropriately referral to other healthcare professionals through the correct detection of referral criteria.
* Record and document of all activities pertaining to the MAS. Intervention: Change Agents - Research Group The research team will provide training, ongoing feedback and support to the FaFas and SeFaFas. The research team will also periodically (at least monthly) hold group meetings by video conference between the research group and all the FaFas and SeFaFas. The agenda will review the progress of the implementation process, as well as resolve any questions related to the study progress. The research group will provide formal reports on the implementation process and patient outcomes which will be discussed at these meetings. Other forms of communication such as emails, telephone calls or WhatsApp messaging will also be available. A research group member has the responsibility of contacting, outside these meetings, as required, FaFas and SeFaFas.

Data: Operational definitions for key process and outcome variables Both implementation and patient consultation process and outcome variables will be measured during the different study stages.

Variables: Implementation indicators

The variables related to the implantation processes and outcomes are:

* Reach of Implementation. The number and percentage of pharmacists at each stage of implementation model i.e. preparation, testing, implementation and initial sustainability will be calculated on a monthly bases extracting data from using the SEFAC eXPERT® IT system
* Fidelity to the Service (degree to which the critical components for the provision of the MAS, i.e., the service is carried out according to how it was standardised). Fidelity will be measured in each pharmacy and will be assessed by the FaFa through role-play and/or other strategies with the pharmacists.
* Integration of the Standardised Service (analysis of the degree of incorporation of the service into the usual practice at the Community Pharmacy): it will be measured through a series of indicators grouped into four dimensions: routinization, evaluation, teamwork and available resources.

Variable: Service indicators Socio-demographic patient characteristics: gender (qualitative dichotomous variables), age (discrete quantitative variable) and physiological state, in the case of pregnancy or lactation.

The variables related to the impact of the MAS are outcome indicators for the clinical and economic and humanistic impact:

* Sociodemographic variables: patient characteristics: gender (qualitative dichotomous variables), age (discrete quantitative variable) and physiological state, in the case of pregnancy or lactation.
* Clinical variables:

  * Type of minor ailment (MA) (five groups), duration of MA (quantitative variable), if it is the first time the patient has suffered this MA, if the MA has already been treated (no/medications/hygienic-dietary measures/food/others).
  * Appropriate referral (dichotomous qualitative variable).
  * Change in the requested treatment (qualitative dichotomous variable).
  * Reason for change: treatment inappropriate for minor ailment, contraindication, incorrect dose, interaction, duplication, inappropriate pharmaceutical form, adverse effect, other drug related problems.
* Humanistic: measure using a visual analogue scale from 0 to 100 for quality of life.

A patient follow up will occur at a maximum of 10 days, depending on the type of consultation. This follow up will be undertaken either through an email or through a face to face meeting the following variables:

* Minor ailment improvement: patient's perception of the resolution of the MA. A Likert scale between 0 (no improvement) and 10 (completely resolved) will be used. In addition, in cases in which there was a complete resolution of the MA, the patient will be asked the number of days elapsed from the consultation in the pharmacy to its complete resolution.
* Repeated consultation for the same minor ailment: in this case the patient will be asked "Did another subsequent consultation for the same minor ailment have to be made?". If so, the patient will be asked the number and type of subsequent consultations i.e a Community Pharmacy, Primary Care physician, or Emergency Services) and the outcome of the consultation (with/without pharmacological treatment, detailing the medication, if any).

Data Analysis Continuous variables will be reported using mean and standard deviation, or median and percentiles depending on the distribution of the variable (the Kolmogorov Smirnov test will be used to assess normality). Categorical variables will be reported using percentages. For the comparison of continuous variables, the T Student's test or the ANOVA test will be carried out if there is a normal distribution, and Kruskal-Wallis otherwise. The comparison of the categorical variables will be carried out using the χ2 test, the Fisher's exact test or Yate's chi-squared test if necessary. To determine the relationship between the dependent variables (appropriate referral, improvement of the minor ailment and subsequent consultation for the same symptom) and the independent variables, logistic regression models will be performed including the variables with statistical significance in the bivariate model. The goodness of fit of the model will be verified using the Hosmer-Lemeshow test. The level of significance will be set at p <0.05. Machine learning and big data techniques are being considered for predictive modelling.

Quality control in data collection The fidelity of the participating pharmacists to the study protocol will be designed using a consensual protocol, and monitored during periodic FaFa visits to the pharmacy, in which the pharmacist's records will be reviewed to ensure that the interventions are carried out according to the protocol for the minor ailment in question. This will allow the FaFas to provide feedback to each participating pharmacist, as a method of continuous quality improvement of their interventions and fidelity to the study.

Data handling The research team will only have access to de-identified data of pharmacists and patients. Data will be extracted form SEFAC eXPERT® IT system by SEFAC staff or contractors.

Informed consent The participating pharmacist will inform patients about the study through a Patient Information Sheet, ensuring that they understand the information before giving their consent. The patient must sign the Informed Consent document (of which they will receive a copy if they should request it), knowing that they may leave the study at any time.

Data confidentiality Privacy protection and the confidential treatment of personal data resulting from the research activity will be guaranteed, in accordance with the provisions of Organic Law 3/2018, of the fifth of December, on the Protection of Personal Data and guarantee of digital rights.

The information will be coded, anonymized and the data will be referenced by randomly assigned numbers for both the published and non-published information. All the information collected will be stored in the repository of the Pharmaceutical Care Research Group of the University of Granada and the Spanish Society of Community Pharmacy (SEFAC), being accessible only to authorized personnel.

Ethical aspects / protection of the participating subjects The study will be carried out following the "Ethical Principles for Medical Research Involving Human Subjects" that are included in the Declaration of Helsinki (Fortaleza, October 2013). The study will be undertaken based on procedures that ensure compliance with the ICH/BPC (International Harmonization Conference) standards of Good Clinical Practice. This study protocol has been approved by the Granada Research Ethics Committee (CEI-Granada) on the fifth of February 2020.

Dissemination Plan The findings obtained after the study will be disseminated through the usual methods of scientific dissemination, including communications to congresses, publications in scientific journals and those of the Pharmaceutical Association, as well as other online or electronic means of dissemination.

Financial Support The study has the financial support of the Spanish Society of Community Pharmacy (SEFAC) and the Pharmaceutical Association of Valencia (MICOF), as well as the participating Pharmacists Associations. Pharmacists participating in this Program will not receive any financial compensation for their participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years or younger if they are accompanied by a responsible adult seeking care i.e. presenting symptoms or requesting a product (direct non-prescription product request) for minor ailments included.
* Patients presenting symptoms or requesting a product for dermatological problems such as acne, bites and stings, cold sore, dermatitis, foot fungi, hyperhidrosis, minor burn, mouth ulcer, rash or soft tissue injury.
* Patients presenting symptoms or requesting a product for gastrointestinal disturbances such as constipation, diarrhoea, flatulence, heartburn or vomiting.
* Patients presenting symptoms or requesting a product for pain-related minor ailments such as dental pain, dysmenorrhea, headache, musculoskeletal pain or sore throat.
* Patients presenting symptoms or requesting a product for upper respiratory tract related ailments such as cold, cough or nasal congestion. Others ailments such as dry eye, haemorrhoids, red eye, sleep problems, stress, temperature, vaginal candidiasis/thrush or varicose veins.

Exclusion Criteria:

• Patients who do not give consent to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20987 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Implementation process of a Minor Ailment Service. | Up to 26 months
  Implementation phases:
  Exploration (number of pharmacists that wish to enrol in the study) Preparation (number of pharmacies that complete the training to provide the Service and record between 1 - 4 consultations per month per pharmacist) Testing (number of pharmacies that record 5 to 10 consultations per month per pharmacist) Implementation (number of pharmacies that perform the MAS on the full number of target patients) Initial sustainability (number of pharmacies that recruit and complete the MAS for the full number of target consultations, 11 or more consultations per month for a further 6 months).
Fidelity of the implementation process of a Minor Ailment Service | Up to 26 months
  Degree to which the critical components for the provision of the Minor Ailment Service are carried out according to how it was standardised. A fifteen-item questionnaire (fidelity questionnaire) is used by the practice change facilitator to evaluate the degree of fidelity for implementing the service for each pharmacist. Each item of the questionnaire uses a 5-item likert scale from very low fidelity to very high fidelity.
Integration of a Minor Ailment Service | Up to 26 months
  Degree of incorporation of the service into the usual practice. A self-administered questionnaire (integration questionnaire) is completed by the pharmacist. Each of the fifteen items of the questionnaire uses a 5-item likert scale from completely disagree (service not integrated in usual practice) to completely agree (service integrated in usual practice).

SECONDARY OUTCOMES:
Appropriate medical referral | Up to 26 months
  Patient referral by the pharmacist made in accordance with the designed protocols, calculated as the proportion of patients appropriately referred divided by the total number of patients.
Rate of modification of direct product request | Up to 26 months
  Treatment requested by the patient modified by the pharmacist due to not approved indication of use for the minor ailment, wrong dose, dosage or formulation. The summary of product characteristics determined by the Spanish Agency was used as the standard.
Symptom resolution | Up to 26 months
  Relief of symptoms measured using a Likert scale from 1 "not at all" to 10 "completely" at 10-day telephone or pharmacy follow-up with interview conducted by the pharmacist.
Reconsultation rate for the same minor ailment | Up to 26 months
  Whenever the patient had to consult again for the same ailment after 10 days of the pharmacist consultation.
Implementation barriers | Up to 26 months
  Measured at the pharmacist-practice change facilitators encounters. The practice change facilitator selects from a list of 62 possible barriers (divided in five domains) those that the pharmacist experiences when implementating the MAS.
Implementation facilitators | Up to 26 months
  Measured at the pharmacist-practice change facilitators encounters. The practice change facilitator selects from a list of 62 possible facilitators (divided in five domains) those that the pharmacist experiences when implementating the MAS.
Interventions used during the implementation | Up to 26 months
  Measured at the pharmacist-practice change facilitators encounters. The practice change facilitator selects from a list of 57 possible interventions (divided in four domains) those used to help the pharmacist to implement the service.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Martínez-Martínez, PhD, Principal Investigator — Pharmaceutical Care Research Group, University of Granada; Jesús C Gómez Martínez, PhD, Study Chair — Spanish Society of Community Pharmacy; Shalom I Benrimoj, PhD, Study Director — Pharmaceutical Care Research Group, University of Granada
Locations (1):
- Spanish Society of Community Pharmacy, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: October 2020-December 2022
Access Criteria: Contact principal investigator

REFERENCES:
- [Background] Allemann SS, van Mil JW, Botermann L, Berger K, Griese N, Hersberger KE. Pharmaceutical care: the PCNE definition 2013. Int J Clin Pharm. 2014 Jun;36(3):544-55. doi: 10.1007/s11096-014-9933-x. Epub 2014 Apr 20. PMID 24748506
- [Background] Moullin JC, Sabater-Hernandez D, Benrimoj SI. Model for the evaluation of implementation programs and professional pharmacy services. Res Social Adm Pharm. 2016 May-Jun;12(3):515-22. doi: 10.1016/j.sapharm.2015.08.003. Epub 2015 Aug 15. PMID 26341944
- [Background] Paudyal V, Hansford D, Cunningham S, Stewart D. Pharmacy assisted patient self care of minor ailments: a chronological review of UK health policy documents and key events 1997-2010. Health Policy. 2011 Aug;101(3):253-9. doi: 10.1016/j.healthpol.2011.05.010. Epub 2011 Jun 15. PMID 21680043
- [Background] Noseworthy J. Minor ailments across Canadian jurisdictions. Can Pharm J (Ott). 2013 Sep;146(5):296-8. doi: 10.1177/1715163513502297. No abstract available. PMID 24137174
- [Background] Hassell K, Whittington Z, Cantrill J, Bates F, Rogers A, Noyce P. Managing demand: transfer of management of self limiting conditions from general practice to community pharmacies. BMJ. 2001 Jul 21;323(7305):146-7. doi: 10.1136/bmj.323.7305.146. No abstract available. PMID 11463686
- [Background] Bojke C, Gravelle H, Hassell K, Whittington Z. Increasing patient choice in primary care: the management of minor ailments. Health Econ. 2004 Jan;13(1):73-86. doi: 10.1002/hec.815. PMID 14724895
- [Background] Baqir W, Learoyd T, Sim A, Todd A. Cost analysis of a community pharmacy 'minor ailment scheme' across three primary care trusts in the North East of England. J Public Health (Oxf). 2011 Dec;33(4):551-5. doi: 10.1093/pubmed/fdr012. Epub 2011 Feb 21. PMID 21339201
- [Background] Pumtong S, Boardman HF, Anderson CW. A multi-method evaluation of the Pharmacy First Minor Ailments scheme. Int J Clin Pharm. 2011 Jun;33(3):573-81. doi: 10.1007/s11096-011-9513-2. Epub 2011 Apr 28. PMID 21526411
- [Background] Paudyal V, Watson MC, Sach T, Porteous T, Bond CM, Wright DJ, Cleland J, Barton G, Holland R. Are pharmacy-based minor ailment schemes a substitute for other service providers? A systematic review. Br J Gen Pract. 2013 Jul;63(612):e472-81. doi: 10.3399/bjgp13X669194. PMID 23834884
- [Background] Watson MC, Ferguson J, Barton GR, Maskrey V, Blyth A, Paudyal V, Bond CM, Holland R, Porteous T, Sach TH, Wright D, Fielding S. A cohort study of influences, health outcomes and costs of patients' health-seeking behaviour for minor ailments from primary and emergency care settings. BMJ Open. 2015 Feb 18;5(2):e006261. doi: 10.1136/bmjopen-2014-006261. PMID 25694456
- [Background] Ocampo CC, Garcia-Cardenas V, Martinez-Martinez F, Benrimoj SI, Amariles P, Gastelurrutia MA. Implementation of medication review with follow-up in a Spanish community pharmacy and its achieved outcomes. Int J Clin Pharm. 2015 Oct;37(5):931-40. doi: 10.1007/s11096-015-0145-9. Epub 2015 Jun 4. PMID 26040837
- [Background] Fuller JM, Saini B, Bosnic-Anticevich S, Garcia Cardenas V, Benrimoj SI, Armour C. Testing evidence routine practice: Using an implementation framework to embed a clinically proven asthma service in Australian community pharmacy. Res Social Adm Pharm. 2017 Sep-Oct;13(5):989-996. doi: 10.1016/j.sapharm.2017.05.019. Epub 2017 May 30. PMID 28583300
- [Background] Garcia-Cardenas V, Benrimoj SI, Ocampo CC, Goyenechea E, Martinez-Martinez F, Gastelurrutia MA. Evaluation of the implementation process and outcomes of a professional pharmacy service in a community pharmacy setting. A case report. Res Social Adm Pharm. 2017 May-Jun;13(3):614-627. doi: 10.1016/j.sapharm.2016.05.048. Epub 2016 Jun 6. PMID 27423785
- [Background] Garcia-Cardenas V, Perez-Escamilla B, Fernandez-Llimos F, Benrimoj SI. The complexity of implementation factors in professional pharmacy services. Res Social Adm Pharm. 2018 May;14(5):498-500. doi: 10.1016/j.sapharm.2017.05.016. Epub 2017 May 29. PMID 28576614
- [Background] Westfall JM, Mold J, Fagnan L. Practice-based research--"Blue Highways" on the NIH roadmap. JAMA. 2007 Jan 24;297(4):403-6. doi: 10.1001/jama.297.4.403. No abstract available. PMID 17244837
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Harvey G, Loftus-Hills A, Rycroft-Malone J, Titchen A, Kitson A, McCormack B, Seers K. Getting evidence into practice: the role and function of facilitation. J Adv Nurs. 2002 Mar;37(6):577-88. doi: 10.1046/j.1365-2648.2002.02126.x. PMID 11879422
- [Background] Baskerville NB, Liddy C, Hogg W. Systematic review and meta-analysis of practice facilitation within primary care settings. Ann Fam Med. 2012 Jan-Feb;10(1):63-74. doi: 10.1370/afm.1312. PMID 22230833
- [Background] Berta W, Cranley L, Dearing JW, Dogherty EJ, Squires JE, Estabrooks CA. Why (we think) facilitation works: insights from organizational learning theory. Implement Sci. 2015 Oct 6;10:141. doi: 10.1186/s13012-015-0323-0. PMID 26443999
- See also: World Health Organization. Self-care in the context of primary health care report of the regional consultation. Bangkok: World Health Organization; 2009. — https://apps.who.int/iris/bitstream/handle/10665/206352/B4301.pdf?sequence=1&isAllowed=y
- See also: Baos Vicente V, Faus Dáder MJ. Protocolos de indicación farmacéutica y criterios de derivación al médico en síntomas menores. Madrid: Fundación Abbott; 2008. — https://digibug.ugr.es/bitstream/handle/10481/33050/ProtocolosIndicacionFarmaceutica.pdf?sequence=1&isAllowed=y
- See also: Foro de Atención Farmacéutica-Farmacia Comunitaria (Foro AF-FC). Guía práctica para los Servicios Profesionales Farmacéuticos Asistenciales en la Farmacia Comunitaria. Madrid: Consejo General de Colegios Oficiales de Farmacéuticos; 2019. — https://www.portalfarma.com/inicio/serviciosprofesionales/forofarmaciacomunitaria/Documents/2019-guia-practica-spfa.pdf
- See also: Real Decreto 109/. Boletín Oficial del Estado núm. 44, de 19/02/2010. — https://www.boe.es/boe/dias/2010/02/19/pdfs/BOE-A-2010-2696.pdf
- See also: Scottish Executive. National Health Service (Scotland) ACT 1978 Health Board additional pharmaceutical services (Minor ailment service) (Scotland) directions. Edinburgh: Scottish Executive; 2006. — https://www.sehd.scot.nhs.uk/pca/PCA2011(P)06.pdf
- See also: Canadian Pharmacists Association. Summary of pharmacists' expanded scope of practice across Canada. Canada: Canadian Pharmacists' Association; 2014. — https://www.pharmacists.ca/pharmacy-in-canada/scope-of-practice-canada/
- See also: NES Pharmacy. Implementation of the minor ailment service introducing the minor ailment service section 1. Scotland: NHS Education for Scotland; 2017 — http://www.nes.scot.nhs.uk/media/426124/1_nes_mas_section1.pdf
- See also: NES Pharmacy. Implementation of the minor ailment service section 5 key steps to implementation of MAS. Scotland: NHS Education for Scotland; 2017 — http://www.nes.scot.nhs.uk/media/426136/5nes_mas_section5.pdf
- See also: Mary Seacole Research Centre. The Pharmacy First Minor Ailments Scheme in Leicester [Internet]. Leicester: Mary Seacole Research Centre; 2011 — https://dora.dmu.ac.uk/bitstream/handle/2086/6214/PHARMAS%20Final_Report_250111_DMU.pdf
- See also: Prats R, Piera V, Pons L, Roig I. Estudio cuantitativo y cualitativo de la indicación farmacéutica en una Farmacia Comunitaria. Pharm Care Esp. 2012;14(1):2-10. — https://www.pharmcareesp.com/index.php/PharmaCARE/article/view/9/9
- See also: Maurandi Guillén MD, Hernández Rex A, Abaurre LabradorR, Arrebola Vargas C, GarcíaDelgado P, Martínez-Martínez F. Satisfacción de los usuarios de Farmacia Comunitaria con un servicio de dispensación pilotado. Ars Pharmaceutica. 2012; 53(2). — https://revistaseug.ugr.es/index.php/ars/article/view/4669/4545
- See also: Eccles MP, Mittman BS. Welcome to Implementation Science. Implementation Science. 2006;1(1). — https://implementationscience.biomedcentral.com/track/pdf/10.1186/1748-5908-1-1.pdf
- See also: Consejo General de Colegios Oficiales de Farmacéuticos, Grupo de Trabajo de Buenas Prácticas. Buenas Prácticas en Farmacia Comunitaria en España, Servicio de Indicación Farmacéutica. Madrid: Consejo General de Colegios Oficiales de Farmacéuticos; 2014. — https://www.portalfarma.com/Profesionales/Buenas-practicas-profesionales/Documents/BBPP-02-ENG-Servicio-Indicacion-Medicamentos.pdf